CLINICAL TRIAL: NCT03229616
Title: Busulfan+ Cyclophosphamide+ Etoposide vs Busulfan+ Cyclophosphamide Conditioning Regimen for Diffuse Large B-cell Lymphoma Undergoing Autologous Hematopoietic Stem Cell Transplantation
Brief Title: BUCY+VP-16 vs BUCY Conditioning Regimen for DLBCL Undergoing Auto-HSCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangzhou First People's Hospital (Other); Zhujiang Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUCY+VP-16 vs BUCY-DLBCL-2017
Record Dates: First submitted 2017-07-23; First posted 2017-07-25 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-07

CONDITIONS: Autologous Hematopoietic Stem Cell Transplantation; Diffuse Large B-cell Lymphoma; Conditioning
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Busulfan; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BUCY+VP-16 (Experimental): For DLBCL patients undergoing auto-HSCT，BUCY+VP-16 conditioning regimen was BU 3.2 mg/kg/day on days -7 and -4；CY 60 mg/kg/day on days -3 and -2; VP-16 15mg/kg/day on days -3 and -2.
  Interventions: Drug: Busulfan (BU); Drug: Cyclophosphamide (CY); Drug: Etoposide (VP-16)
- BUCY (Active Comparator): For DLBCL patients undergoing auto-HSCT，BUCY conditioning regimen was BU 3.2 mg/kg/day on days -7 and -4；CY 60 mg/kg/day on days -3 and -2.
  Interventions: Drug: Busulfan (BU); Drug: Cyclophosphamide (CY)

INTERVENTIONS:
Drug: Busulfan (BU) — Busulfan was administered at 3.2 mg/kg/day on days -7 to -4.
Drug: Cyclophosphamide (CY) — Cyclophosphamide was administered at 60 mg/kg/day on days -3 to -2.
Drug: Etoposide (VP-16) — Etoposide was administered at 15 mg/kg/day on days -3 to -2.
  Arms: BUCY+VP-16

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of BUCY+VP-16 and BUCY myeloablative conditioning regimens in diffuse large B-cell lymphoma undergoing autologous hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Autologous hematopoietic stem cell transplantation (Auto-HSCT) is an effective therapy for diffuse large B-cell lymphoma (DLBCL).BuCY conditioning regimen is a conventional scheme for DLBCL patients undergoing auto-HSCT, but it has a high relapse rate. Etoposide (VP-16) is extensively used in chemotherapy regimen for refractory/relapsed lymphoma. Whether addition of VP-16 could reduce the relapse rate remains unclear.In this study, the safety and efficacy of BUCY+VP-16 and BUCY myeloablative conditioning regimens in DLBCL undergoing auto-HSCT are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diffuse large B-cell lymphoma patients
* Achieving CR or PR after four cycles of chemotherapy, then mobilizing and collecting of peripheral blood stem cells and receiving one cycle of chemotherapy

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
relapse rate | 2 year
  relapse rate

SECONDARY OUTCOMES:
DFS | 2 year
  disease-free survival (DFS)
OS | 2 year
  overall survival (OS)
TRM | 2 year
  transplant-related mortality (TRM)

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided